CLINICAL TRIAL: NCT04281940
Title: Chordal Repair for Transcatheter Mitral Valve Repair (TMVr)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pipeline Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0001
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Degenerative Mitral Valve Disease; Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Permanent Implant (Experimental): Insertion of the Chordal Repair System tethering the mitral leaflets to the left ventricle.
  Interventions: Device: Transcatheter implantation of chordal repair system

INTERVENTIONS:
Device: Transcatheter implantation of chordal repair system — Implantation of anchor via transcatheter delivery system to delivery chordal repair system tethering the mitral leaflets to the ventricle

SUMMARY:
A multi-center evaluation of the Pipeline chordal repair system for treatment of clinically significant mitral regurgitation in subjects determined appropriate for mitral valve repair.

DETAILED DESCRIPTION:
The proposed study is a prospective, multi-center, interventional investigation enrolling up to 30 subjects in multiple sites in Latin America and Eastern Europe.

The primary objective of this study is to collect preliminary information on the performance and safety of the Pipeline Chordal Repair System in percutaneous reduction of significant mitral regurgitation (MR ≥ moderate) due to primary abnormality of the mitral apparatus [degenerative MR].

ELIGIBILITY:
Inclusion Criteria:

* Presence of moderate to severe Mitral regurgitation as read on an echocardiographic study performed within 60 days prior to procedure.
* Estimated post-ePTFE chordae tendineae implantation coaptation surface is adequate in the judgment of the operating physician and the patient eligibility committee.
* Degenerative mitral valve disease.
* Patients who have been evaluated and no contraindication has been found for open heart surgery OR candidates for mitral valve surgery who, according to current guidelines, are at elevated surgical risk AND for whom transcatheter therapy is deemed more appropriate than open heart surgery in the judgement of the Site Heart Team.

Exclusion Criteria:

* Untreated clinically significant coronary artery disease requiring revascularization
* Creatine Kinase-MB (CK-MB) obtained within prior 14 days > local laboratory Upper Limit of Normal (ULN)
* Age <30/40 or > 85 years
* Presence of any of the following:
* Estimated pulmonary artery systolic pressure (PASP) > 70 mmHg assessed by site based on echocardiography or right heart catheterization
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, ischemic or non-ischemic Functional mitral regurgitation or any other structural heart disease causing heart failure
* Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis)
* Hemodynamic instability requiring inotropic support or mechanical heart assistance
* Hemodynamic instability defined as systolic pressure < 90 mmHg with or without afterload reduction, cardiogenic shock or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device
* Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction
* Left Ventricular Ejection Fraction (LVEF) is < 30% (within 90 days prior to subject enrollment, assessed by the site using any one of the following methods: echocardiography, contrast left ventriculography, gated blood pool scan or cardiac magnetic resonance imaging (MRI))
* Mitral annular diameter >45mm in any dimension. Left Ventricular End Diastolic Diameter (LVEDD) > 65mm. Left Ventricular End Systolic Dimension (LVESD) > 55 mm assessed by site based on a transthoracic echocardiographic (TTE) obtained within 90 days prior to subject enrollment
* Coronary artery bypass grafting (CABG) within 30 days prior to subject's consent
* Percutaneous coronary intervention within 30 days prior to subject's consent
* Tricuspid valve disease requiring surgery
* Aortic valve disease requiring surgery or TAVI
* Carotid surgery within 30 days prior to subject's consent
* Implant of any Cardiac Resynchronization Therapy (CRT) or Cardiac Resynchronization Therapy with cardioverter-defibrillator (CRT-D) within the last 30 days prior to subject's consent
* Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months
* Prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure
* Status 1 heart transplant or prior orthotopic heart transplantation
* Chronic Kidney Disease with a baseline serum creatinine > 1.5mg/dL
* Chronic Steroid Therapy
* Cerebrovascular accident within 30 days prior to subject's consent
* Severe symptomatic carotid stenosis (> 70 % via ultrasound)
* Life expectancy < 12 months due to non-cardiac conditions
* Active infections requiring current antibiotic therapy
* Pregnant or planning pregnancy within next 12 months
* Currently participating in an investigational drug or another device study
* Severe organic lesions with mitral chords retraction, severely fibrotic and immobile leaflets, severely deformed subvalvular apparatus
* Evolving endocarditis or active endocarditis in the last 3 months
* Heavily calcified or dilated annulus or leaflets, mitral valve stenosis
* Congenital malformation with limited valvular tissue
* Patient requires mitral valve replacement
* Previously implanted prosthetic mitral valve or annuloplasty ring/band
* Evidence of LV or LA thrombus, vegetation or mass
* Severe tricuspid regurgitation or severe RV dysfunction
* Condition that prevents transfemoral access
* Anatomical ineligibility to the investigational device
* Known hypersensitivity or contraindication to procedural, post procedural medication (e.g., contrast solution, anticoagulation therapy) or hypersensitivity to nickel or titanium

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Safety at 30 days: freedom from death or intervention resulting from valve dysfunction or the implant procedure at 30 days. | Procedure through 30 days post procedure
  Primary Safety
Freedom from device-related Major Adverse Events (MAE), defined as a combined clinical endpoint of death, reoperation for failed surgical repair or replacement, non-elective cardiovascular surgery for adverse events, stroke or renal failure | Procedure through 30 days post procedure
  Primary Safety
Technical successful transcatheter implantation of the Chordal Repair System tethering the mitral leaflets to the ventricle | Procedure
  Technical Success
Procedural success defined as the successful implant of the device resulting in MR severity of < moderate at 30 days as confirmed by echocardiography. | Procedure through 30 days post procedure
  Procedural Success

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Principal Investigator
Locations (4):
- Israeli-Georgian Medical Research Clinic Healthycore, LTD, Tbilisi, Georgia
- Sanatorio Italiano, Asunción, Paraguay
- Serbia (2):
  - Institute for Cardiovascular Diseases Dedinje, Belgrade
  - Institute for Cardiovascular Diseases Vojvodina, Kamenitz

IPD SHARING:
Plan to Share IPD: No